CLINICAL TRIAL: NCT03146507
Title: Doppler Echocardiography Assessment of Cardiac Sparing Effect in Fetal Hypoxia
Brief Title: Assessment of Cardiac Sparing in Fetal Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sief el eslam Ahmed Ali, Principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AU03
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Fetal Hypoxia
MeSH Terms: conditions — Fetal Hypoxia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal pregnant women at 32-34 weeks group (Other)
  Interventions: Radiation: Ultrasound; Radiation: Doppler ultrasound; Radiation: Fetal echocardiography
- Intrauterine growth restriction at 32-34 weeks group (Other)
  Interventions: Radiation: Ultrasound; Radiation: Doppler ultrasound; Radiation: Fetal echocardiography

INTERVENTIONS:
Radiation: Ultrasound — ultrasound assessment of gestational age, amniotic fluid index, and fetal weight
Radiation: Doppler ultrasound — Umbilical artery and Middle cerebral artery Doppler blood flow assesment
Radiation: Fetal echocardiography — The cardiac output (ratio between right side cardiac outputs to left side cardiac output) was calculated

SUMMARY:
The fetal heart plays a central role in the adaptive mechanisms for hypoxemia and placental insufficiency. Longitudinal data on the hemodynamic sequence of the natural history of fetal growth restriction show that the umbilical artery and middle cerebral artery are the first variables to become abnormal . These arterial Doppler abnormalities are followed by abnormalities in the right cardiac diastolic indices, followed by the right cardiac systolic indices, and finally by both left diastolic and systolic cardiac indices .

Preserving the left systolic function as the last variable to become abnormal ensures an adequate left ventricular output , which supplies the cerebral and coronary circulations.This defence is contingent on the fetal cardiovascular system, which in late gestation adopts strategies to decrease oxygen consumption and redistribute the cardiac output away from peripheral vascular beds and towards essential circulations, such as those perfusing the brain.

Adding cardiac Doppler may improve management of the IUGR fetus(intrauterine growth retardation), Doppler ultrasound is valuable in defining the degree of cardiovascular compromise in at-risk pregnancies. The severity of fetal blood flow redistribution shows the degree of fetal adaptation and provides information on how long the pregnancy can be continued safely.

The aime of the study is assessment of cardiac output redistribution in fetal hypoxia by estimating relative right to left side cardiac output wich reflect cardiac sparing in (IUGR).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-35 years.
2. Women with BMI from 20-30 kg/m2.
3. Pregnant women in singleton fetuses from 32 to 34 weeks gestation.
4. Women with late fetal growth restriction fetuses. It refers to an estimated fetal weight or abdominal circumference <10th centile. Those women had increased the resistant index (RI) in umbilical arteries above the 95th percentile at the time of recruitment (case group).
5. Normal pregnant women (control group).

Exclusion Criteria:

1. Women with estimated fetal weight below the 5th or 3rd percentile.
2. Women with premature pre-labor rupture of membranes.
3. Women with antepartum hemorrhage
4. Women with fetal congenital anomalies.
5. Women with absent or reversed diastolic flow in the umbilical artery at the time of recruitment.
6. Women with preeclampsia or on anti-coagulant thereby.
7. Women who refused to participate in our study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The relative cardiac output ratio (ratio between right side cardiac outputs to left side) cardiac output) at 32-34 weeks. | 1 month

SECONDARY OUTCOMES:
The relative cardiac output ratio at 34-36 weeks. | 1 month
The pulsatility index in the umbilical artery and middle cerebral artery at 32-34 weeks | 1 month
The pulsatility index in the umbilical artery and middle cerebral artery at 34-36 weeks | 1 month
Middle cerebral artery pulsatility index to umbilical artery pulsatility index ratio | 15 minutes
Time of delivery (weeks) | 7 weeks
Birth weight (grams) | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Fetal Cair Unit - Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes